CLINICAL TRIAL: NCT01258296
Title: Postoperative Pain Control With Fentanyl Patch in Patients Undergoing Mastectomy and TRAM or DIEP Flap Reconstruction
Acronym: Fentanyl Patch
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Laura Esserman, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCSF-04804
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2010-12

CONDITIONS: Postoperative Pain After Breast Reconstruction With Abdominal Flap
Keywords: Postoperative pain; Breast reconstruction; Abdominal flap breast reconstruction
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active fentanyl patch (Active Comparator): 25 mcg/hr fentanyl patch
  Interventions: Drug: Fentanyl
- Placebo patch (Placebo Comparator): Inactive patch that resembles treatment patch but contains no drug
  Interventions: Drug: Inactive patch

INTERVENTIONS:
Drug: Fentanyl — 25 mcg/hr transdermal patch
  Arms: Active fentanyl patch
Drug: Inactive patch — placebo patch (no drug)
  Arms: Placebo patch

SUMMARY:
The aim of this randomized, double-blind controlled trial is to determine the efficacy of transdermal fentanyl for the management of early postoperative pain in women undergoing mastectomy followed by immediate TRAM or DIEP flap reconstruction. We will examine whether the use of the fentanyl patch as a bridge between epidural and oral analgesia will improve overall pain relief compared to placebo patch. We further propose to study whether the fentanyl patch is associated with improved ability to sleep, patient satisfaction, and functional capacity at one week, and whether it is associated with different side effects than standard therapy without the patch. Following informed consent, patients will undergo mastectomy and reconstruction, and receive epidural fentanyl for initial postoperative analgesia. Patients will be randomized to active (25 mcg/hr Duragesic) or placebo patches on postoperative day three, and the epidural will be weaned over the next 12 hours. Pain intensity scores and relief from pain will be assessed every day while in the hospital and oral and IV opioid use recorded. Patients will be discharged to home with a supply of 2 patches and oral medication, and will be asked to fill out a daily pain and medication log.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing breast reconstruction with abdominal flap
* Provided written, informed consent

Exclusion Criteria:

* Karnofsky performance status ≥80%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Opioid analgesic use | 10-20 days
  Daily opioid use on immediate postoperative days while wearing patch

SECONDARY OUTCOMES:
Pain intensity | 10-20 days
  Daily measure of pain intensity on 0-10 numeric rating scale on postoperative days
Relief from pain | 10-20 days
  Daily measure of relief provided by pain medications on 0-100% scale on postoperative days
Adverse event questionnaire | 10-20 days
  Daily measurement of headache, itching, nausea, vomiting, constipation, difficulty urinating, drowsiness, lightheadedness, indigestion
Functional assessment questionnaire | 10-20 days
  Daily measure of how surgical pain has interfered with general activity, mood, walking ability, sleep, brushing teeth, interactions with other people and enjoyment of life on a 0-10 scale on postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Laura Esserman, MD, Principal Investigator — University of California, San Francisco; Laura Petrillo, BA, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States